CLINICAL TRIAL: NCT04733183
Title: A Randomized Study to Investigate the Efficacy and Safety of the Tumor-targeting Human Antibody-cytokine Fusion Protein L19TNF in Previously Treated Patients with Advanced Stage or Metastatic Soft-tissue Sarcoma
Brief Title: Efficacy and Safety of L19TNF in Previously Treated Patients with Advanced Stage or Metastatic Soft-tissue Sarcoma
Acronym: FLASH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFSARC-03/18
Record Dates: First submitted 2021-01-22; First posted 2021-02-01 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Dacarbazine

STUDY DESIGN:
Intervention Model Description: Safety Run in: Six (6) Patients will be treated with 1000 or 850 mg/m2 dacarbazine (DTIC) on Day 1 every three weeks plus 13 µg/kg L19TNF on Days 1, 3 and 5 every three weeks to test for safety of the combination as evaluated by an independent Data Safety Monitoring Board (DSMB).
  Tumor Activity Evaluation Part Arm 1: Patients will receive DTIC on Day 1 and L19TNF on Days 1, 3 and 5 every 3 weeks.
  Arm 2: Patients will receive DTIC on Day 1 every 3 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm1: DTIC + L19TNF (Experimental): Patients will receive Dacarbazine (DTIC) on Day 1 and L19TNF on Days 1, 3 and 5 every 21 days.
  Interventions: Drug: Dacarbazine; Drug: onfekafusp alfa
- Arm 2: DTIC (Active Comparator): Patients will receive Dacarbazine (DTIC) on Day 1 every 21-day cycle .
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Dacarbazine — Dacarbazine (DTIC), 1000 mg/m2 or 850 mg/m2 on Day 1 of every 21-day cycle (based on results and DSMB evaluation in the safety run-in part of the study)
  Other Names: DTIC
Drug: onfekafusp alfa — L19TNF, 13 μg/kg, on Day 1, 3, and 5 of every 21-day cycle for a maximum of 6 induction cycles. Patients experiencing apparent or real benefit with minimal or acceptable toxicity from the first 6 cycles of treatment, can receive, at investigator's discretion, maintenance treatment of 13 μg/kg, on Day 1 every 21-day
  Other Names: L19TNF
  Arms: Arm1: DTIC + L19TNF

SUMMARY:
Open label, randomized, controlled phase II study preceded by a safety run-in part in subjects with advanced or metastatic soft-tissue sarcoma.

DETAILED DESCRIPTION:
Open label, randomized, controlled phase II study preceded by a safety run-in part in subjects with advanced or metastatic soft-tissue sarcoma.

* Safety Run-in Part: Six (6) patients will be treated with 1000 mg/m2 dacarbazine (DTIC) on Day 1 every 3 weeks plus 13 µg/kg L19TNF on Days 1, 3 and 5 every 3 weeks to test for safety of the combination. Should unacceptable toxicities occur in ≥ 2 patients during an observation period from Day 1 to Day 21 (first cycle), enrollment will be stopped at this dose level and 6 patients will be treated sequentially with DTIC at 850 mg/m2 on Day 1 every 3 weeks plus 13 µg/kg L19TNF on Days 1, 3 and 5 every 3 weeks.
* Tumor Activity Evaluation Part

Approximately 86 patients will be enrolled and parallel assigned in a 1:1 fashion to one of two different arms, as follows:

* Arm 1: Patients will receive DTIC on Day 1 every 3 weeks plus L19TNF on Days 1, 3 and 5 every 3 weeks.
* Arm 2: Patients will receive DTIC on Day 1 every 3 weeks. During the conduct of the study, detailed safety parameters will be routinely reviewed by the DSMB.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 80 years of age.
2. Histologically or cytologically confirmed advanced unresectable or metastatic soft tissue sarcoma (STS), Grade 2 - 3 according to the FNLCC grading system. Participants with bone sarcomas including Ewing sarcoma, Kaposi's sarcoma and gastrointestinal stromal tumors (GIST) will be excluded.
3. Subjects who received at least two prior systemic therapies (e.g., anthracyclines, taxanes, ifosfamide, gemcitabine, trabectedin, pazopanib, eribulin) for advanced or metastatic disease including at least one prior therapy based on anthracyclines as monotherapy or in combination. Neoadjuvant and adjuvant therapies can be considered as a prior line of treatment if the time to recurrence from completion of treatment was ≤ 12 months. Previous therapy with anthracyclines is not compulsory in situations of contraindications to this class of drugs. All previous therapies must have completed ≥ 3 weeks (21 days) prior to study treatment start.
4. Evidence of disease progression after prior line of therapy for advanced or metastatic disease.
5. Patients must have at least one unidimensionally measurable lesion by computed tomography as defined by RECIST criteria v.1.1. If only one lesion is present at screening this lesion should not have been irradiated during previous treatments.
6. Life expectancy of at least 3 months in the judgment of the investigator.
7. ECOG ≤ 2.
8. Documented negative test for HIV-HBV-HCV. For HBV serology: the determination of HBsAg and anti-HBcAg-Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required. For HCV: HCV-RNA or HCV antibody test. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
9. Female patients: negative serum pregnancy test at screening for women of childbearing potential (WOCBP)*. WOCBP must agree to use, from the screening to six months following the last study administration of L19TNF and/or DTIC, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence. Male patients: Male subjects able to father children must agree to use two acceptable methods of contraception throughout the study from the screening to six months following the last administration of L19TNF and/or DTIC (e.g. condom with spermicidal gel). Double-barrier contraception is required.
10. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
11. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

    * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

Exclusion Criteria:

1. Anti-cancer treatment with radiation therapy (with the exception of radiation of single lesions for palliative reasons, e.g. pain management which then are not taken as indicator lesions for iRECIST response), chemotherapy, targeted therapies, immunotherapy, hormones or other antitumor therapies within 3 weeks prior to study treatment start.
2. Subjects who participated in an investigational drug or device study within 3 weeks prior to study treatment start.
3. Previous treatment with TNF or L19TNF or DTIC.
4. Known history of allergy to intravenously administered human proteins/peptides/antibodies and any other constituent of the product.
5. Absolute neutrophil count (ANC) < 1.5 x 109/L, platelets < 100 x 109/L and hemoglobin (Hb) < 9.0 g/dl, with the exception of values lower than these due to cytologically or histologically proven marrow metastasis, which will not constitute exclusion criteria.
6. Chronically impaired renal function as expressed by creatinine clearance < 60 mL/min or serum creatinine > 1.5 ULN.
7. Inadequate liver function (ALT or AST ≥ 3 x ULN or ALP or GGT ≥ 2.5 x ULN, or total bilirubin ≥ 1.5 x ULN). For patients with metastatic lesions in the liver ALT, AST, GGT or ALP ≥ 5 x ULN.
8. Any severe concomitant condition which in the opinion of investigators makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
9. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
10. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
11. Clinically significant cardiac arrhythmias.
12. Abnormalities observed during baseline ECG and echocardiogram investigations that are considered as clinically significant by the investigator.
13. Uncontrolled hypertension.
14. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
15. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
16. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
17. Pregnancy or breast-feeding.
18. Requirement of chronic administration of corticosteroids or other immunosuppressant drugs. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
19. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
20. Known active or latent tuberculosis (TB).
21. Concurrent malignancies other than soft-tissue sarcoma, unless the patient has been disease-free for at least 2 years.
22. Serious, non-healing wound, ulcer or bone fracture.
23. Allergy to study medication or excipients in study medication.
24. Deep vein thrombosis, pulmonary embolism or other acute vascular events within 6 months
25. Anticoagulation therapy with P2Y12 antagonists (e.g., clopidogrel, ticagrelor) and vitamin K antagonists (e.g., phenprocoumon, warfarin).
26. Concurrent use of other anti-cancer treatments or agents other than study medication.
27. Protected adults (i.e., persons referred to as adults who are under legal protection measure or unable to express their consent) or persons under the protection of justice.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | The PFS rate will be assessed at 3 months.
  Progression-free survival (PFS) in according to RECIST v.1.1. The duration is defined beginning from randomization to progression or death from any cause.
Progression-free survival (PFS) | The PFS rate will be assessed at 6 months.
  Progression-free survival (PFS) in according to RECIST v.1.1. The duration is defined beginning from randomization to progression or death from any cause.
Progression-free survival (PFS) | The PFS rate will be assessed at 9 months.
  Progression-free survival (PFS) in according to RECIST v.1.1. The duration is defined beginning from randomization to progression or death from any cause.
Progression-free survival (PFS) | The PFS rate will be assessed at 12 months.
  Progression-free survival (PFS) in according to RECIST v.1.1. The duration is defined beginning from randomization to progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | The OS will be calculated at 12, 18, 24 and 36 months.
  Overall Survival (OS) will be assessed for all randomized patients. The duration is defined beginning from randomization to death from any cause.
Objective response rate (ORR) | The ORR rate will be assessed at 3, 6, 9, 12 months.
  Objective response rate (ORR, consisting of CR plus PR; only the non-irradiated lesions are measured) according to RECIST v.1.1 between arms.
Objective Response Rate (ORR) | The ORR rate will be assessed at 3, 6, 9, 12 months.
  Objective Response Rate (ORR, consisting of iCR plus iPR; only the non-irradiated lesions are measured) according to iRECIST in Arm1.
Adverse Events | Time Frame: From week 1 up to week 52
  Number of patients with adverse events (AEs) assessed on CTCAE v.4.03
HAFA assessment | At day 1 of week 1 and week 2; at day 1 from week 4 up to week 18; at week 22 (EoT)
  Assessment of the formation of human anti-fusion protein antibodies (HAFA) against L19TNF.
Quality of life (HRQol) | EORTC Quality of Life Questionnaire C30 will be assessed baseline at 3, 6, 9 and 12 months and EOT visit (if not done already within 4 weeks prior)
  Quality of life of L19TNF in combination with DTIC compared to DTIC alone as Health-related Quality of life (HRQol)

CONTACTS AND LOCATIONS:
Locations (23):
- France (8):
  - Hopital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut régional du Cancer de Montepellier - ICM Val d'Aurelle, Montpellier
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Münster University Hospital, Münster, Münster
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Helios Klinikum Berlin- Buch, Berlin
  - Klinik rechts der Isar, TU München, München
- Italy (4):
  - IRCCS - Istituto Ortopedico Rizzoli, Bologna
  - IRCCS Fondazione del Piemonte per l'Oncologia Istituto per la Ricerca e la Cura del Cancro di Candiolo, Candiolo
  - AOU San Luigi Gonzaga, Orbassano
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Poland (2):
  - Szpital Pomorski Im. PCK, Gdynia
  - Maria Sklodowska Curie National Research Institute of Oncology, Warsaw
- Spain (5):
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No